CLINICAL TRIAL: NCT03918681
Title: Gait Retraining Enhances Athletes' Technique: GREAT After Anterior Cruciate Ligament Reconstruction
Brief Title: Gait Retraining Enhances Athletes' Technique
Acronym: GREAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We terminated the study due to covid 19 difficulties.
Sponsor: Keller Army Community Hospital (U.S. Federal Agency)
Collaborators: Telemedicine & Advanced Technology Research Center (Other)
Responsible Party: Principal Investigator, Jamie Morris, Director & Associate Professor, Keller Army Community Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19KACH001
Record Dates: First submitted 2019-02-15; First posted 2019-04-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament Injury; Knee Osteoarthritis
Keywords: Running; Gait Retraining; Return to Run; ACLR; Loading
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis, Knee | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: pre-test, post-test, single-blind randomized controlled trial study design
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors will be blind to treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The experimental group participants (approximately 20 participants) will receive, a standard graduated return-to-run program, a 4-week lower-extremity exercise program, and an activity log to track exercise progress. Participants will be instructed to follow-up with their research physical therapist once a week for the first 4 weeks and then every other week until the run progression is completed. During follow-ups experimental group participants will receive gait retraining cues to transition to a NRFS running pattern.
  Interventions: Other: Therapeutic Intervention
- Control Group (No Intervention): The control group participants (approximately 20 participants) will receive, a standard graduated return-to-run program, a 4-week lower-extremity exercise program, and an activity log to track exercise progress. Participants will be instructed to follow-up with their research physical therapist once a week for the first 4 weeks and then every other week until the run progression is completed. During follow-ups control group participants will not receive any gait retraining cues and will only be instructed on standard of care return to run metrics to include volume, load, and duration of running.

INTERVENTIONS:
Other: Therapeutic Intervention — Instruction for all participants in the experimental group will begin with transitioning foot strike pattern from a rearfoot strike to a non-rearfoot strike running pattern (NRFS) and increasing preferred step rate by 5-10%. Each participant program thereafter will be progressed individually according to the clinical investigators follow up assessments of running mechanics and participant pain and function with running. Intervention gait retraining sessions will include drills for reinforcement to include soft landing single leg bounding, adequate time to practice, and pre-class and post-class video assessment with feedback.
  Other Names: Gait Retraining
  Arms: Intervention Group

SUMMARY:
The participant population for this study will be a convenience sample of 40 active duty soldiers and cadets at West Point, New York (NY) who are recovering from anterior cruciate ligament reconstruction (ACLR) and are cleared to return to run by their medical provider. Two groups will be utilized in this pre-test, post-test, single-blind randomized controlled trial study design. The purpose of this study is to determine if patients recovering from ACLR benefit from running gait retraining to adopt a forefoot strike pattern and 5-10% increase in step rate when compared to a traditional walk to run program.

DETAILED DESCRIPTION:
The participant population for this study will be a convenience sample of 40 active duty soldiers and cadets at West Point, NY who are recovering from Anterior Cruciate Ligament Reconstruction (ACLR) and are cleared to return to run by their medical provider. Two groups will be utilized in this repeated measures, single-blind, randomized controlled trial study design. The purpose of this study is to determine if patients recovering from ACLR benefit from running gait retraining when compared to a traditional walk-to-run program. Patient reported outcome measures, running kinetic data and running kinematic data, along with biomarkers of cartilage turnover and clinical outcomes will be assessed in two groups of post-operative ACLR patients. All participants, regardless of group, will be instructed in a 4-week home exercise program to ensure runners have adequate strength prior to returning to full running activities. They will be provided an instructional handout and compliance log at the date of their initial running biomechanical assessment. The home exercise program will consist of exercises focused on stretching and strengthening of the hip, knee, calf and foot musculature. One group will receive technology assisted clinician guided gait retraining to reduce lower extremity loading parameters (intervention) while the control group will return to running with a traditional return to run program (control). Regardless of group, all runners will have their running form and foot strike pattern analyzed using an instrumented treadmill and high-speed motion capture initially, at the pre-intervention, post-intervention, and follow-up time point. During the intervention period, regardless of group, all runners will complete in-clinic follow-ups with their study assigned medical provider. During these visits the control group will only receive standard run program feedback. During these visits the intervention group will receive technology-guided clinician-assisted gait retraining cues to reduce ground reaction forces during running. Kinetic data, kinematic data, and perceived running pain and running function will be collected at the pre-intervention, post-intervention and follow-up timepoints to include average vertical loading rate (AVLR), AVLR symmetry, impulse, foot strike pattern (FSP), contact time, step length, step rate, Visual Analog Scale for Running Pain during running, Visual Analog Scale for Running Pain worst pain, Visual Analog Scale for Running Pain during after running, Single Assessment Numeric Evaluation, Knee Injury and Osteoarthritis Outcome Score (KOOS), and University of Wisconsin Running and Recovery Index (UWRI). Biological samples will be collected from all runners regardless of group at the pre-intervention time point and the post-intervention timepoint. Biological samples will be tested using ELISA for several biomarkers of interest and the concentration of these biomarkers will be compared within and between groups over time. A pan-omics (e.g. metabolomics, proteomics, and transcriptomics) approach will be used to test for novel biomarkers that will also compare within and between groups over time. Our military service members are at greater risk of ACL injury, greater risk of early onset knee Osteoarthritis (OA), and are required to maintain high levels of fitness to remain in the military. It is therefore clinically important to identify interventions to improve patient reported outcomes, return to duty rates, and reduce lower extremity loading parameters in military service members returning to run after ACLR.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give informed consent
2. Between 18-50 years of age
3. Active duty Soldier or cadet
4. History of Anterior Cruciate Ligament Reconstruction in the last 18 months
5. Cleared to return to run by their Department of Defense medical provider (primary care physician, orthopedic surgeon, physical therapist, or athletic trainer)
6. Ability to perform 20 unassisted single leg heel raises bilaterally
7. Ability to perform 10 pain-free, symmetrical, single-leg squats to between 45-60 degrees bilaterally
8. Ability to perform 20 pain-free single leg hops in place bilaterally

Exclusion Criteria:

1. Currently on an Army running limiting profile
2. Concomitant Posterior Cruciate Ligament or Lateral Cruciate Ligament injury
3. Concomitant meniscectomy >50%
4. History of inflammatory arthritis or gout
5. History of ACL injury to either knee
6. History of major lower-extremity joint injury and/or surgery
7. Known pregnancy currently or in the previous 6 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) During Running Pain | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  VAS, measures self-reported pain, scored on a 0-10 scale with 0 being no pain and 10 being worst pain imaginable.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  Subjective Knee Evaluation Form

SECONDARY OUTCOMES:
University of Wisconsin Running and Recovery Index (UWRI) | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  UWRI, scored on a scale from 0-36 with 36 equaling completion of running function and a score of 0 equating to inability to run.
CPII Serum Biomarker Concentration | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  Blood specimen biomarker associated with knee osteoarthritis and cartilage/bone turnover.
C1 Serum Biomarker Concentration | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  Blood specimen biomarker associated with knee osteoarthritis and cartilage/bone turnover.
2C Serum Biomarker Concentration | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  Blood specimen biomarker associated with knee osteoarthritis and cartilage/bone turnover.
C2C Serum Biomarker Concentration | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  Blood specimen biomarker associated with knee osteoarthritis and cartilage/bone turnover.
CTX-1 Serum Biomarker Concentration | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  Blood specimen biomarker associated with knee osteoarthritis and cartilage/bone turnover.
NTX Serum Biomarker Concentration | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  Blood specimen biomarker associated with knee osteoarthritis and cartilage/bone turnover.
Average Vertical Loading Rate (AVLR) | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  A vertical ground reaction force measure that indicates how quickly force is being applied to the body.

OTHER OUTCOMES:
Patient Specific Functional Scale (PSFS) | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  PSFS, scored on a 0-10 scale with six pre-filled items: walking, running on level ground less than 2 miles, running uphill, running downhill, running on level ground greater than 2 miles, and hopping/jumping).
Single Assessment Numeric Evaluation (SANE) | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  SANE, scored on a 0-100% scale with 100% equaling completion of function
Peak Vertical Ground Reaction Force | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  A vertical ground reaction force measure that indicates how the peak force applied to the body.
Braking Force | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  A vertical ground reaction force measure that indicates the amount of anterior force applied to the body.
Vertical Center of Mass Displacement | Change from Pre-Intervention (Initial) to Post-Intervention (up to 10 weeks). Change from Pre-Intervention (Initial) to Follow-Up (Up to 15 weeks)
  The difference between the highest vertical and lowest vertical point achieved during a running stride.

CONTACTS AND LOCATIONS:
Overall Officials: Erin M Miller, MS, ABD, Principal Investigator — Keller Army Community Hospital
Locations (1):
- Keller Army Community Hospital, West Point, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT03918681/ICF_000.pdf